CLINICAL TRIAL: NCT02314572
Title: Evaluation of the Visual Acuity After the Implantation of a ReSTOR +2.5 Diopters Intraocular Lens (ReSTOR SV25T0) in the Distance Dominant Eye, in Combination With a +3.0 Diopters ReSTOR Intraocular Lens (ReSTOR SN6AD1) in the Fellow Eye.
Brief Title: Visual Acuity After the Combined Binocular Implantation of +2.5 Diopters and +3.0 Diopters ReSTOR Multifocal Intraocular Lenses.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, PD Dr. med. Eckart Bertelmann, managing senior physician, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA1/124/13
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Cataract
Keywords: Multifocal Intraocular Lens; Binocular Trifocality; Cataract Surgery; Spectacle Independence; Intermediate Vision; Photopic Vision; Mesopic Vision; Scotopic Vision; Binocular Vision
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Other)
  Interventions: Device: Binocular cataract surgery with phacoemulsification and implantation of multifocal intraocular lenses

INTERVENTIONS:
Device: Binocular cataract surgery with phacoemulsification and implantation of multifocal intraocular lenses — Binocular implantation of the combination of AcrySof® IQ ReSTOR® multifocal intraocular lenses with an addition of +2.5 D in the distance-dominant eye and +3.0 D in the fellow eye.
  Other Names: AcrySof® IQ ReSTOR® multifocal intraocular lenses with an addition of +2.5 D (SV25-type) and +3.0 D (SN6A-type) are used.

SUMMARY:
The objective of this study is to assess the visual outcome after the combined binocular implantation of +2.5 D and +3.0 D apodized diffractive multifocal intraocular lenses.

DETAILED DESCRIPTION:
Bifocal multifocal intraocular lenses (MIOL) are effective in achieving good uncorrected visual acuities in the distance and the near. However, the intermediate vision is of increasing relevance for everyday's life. Several multifocal intraocular lenses have been developed to improvement intermediate vision. Nonetheless, those systems still possess adverse photic effects and do not garantuee spectacle independence. Therefore, the combination of a lower-addition bifocal intraocular lense in the distance-dominant eye with a higher-addition bifocal intraocular lense in the fellow-eye might be a promising approach to address these drawbacks of current binocular and trifocal intraocular lenses.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant cataract
* endothelial cell count: patients aged 18-75 years: > 1000 cells/mm2; patients > 75 years: > 750 cells/mm2
* absence of vision-limiting corneal or retinal comorbidities
* capability to understand the informed consent

Exclusion Criteria:

* expected postoperative astigmatism > 0.75 diopters
* irregular astigmatism
* dilated pupil diameter < 3 mm
* corneal and fundus abnormalities that might cause visual impairments
* inability to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Visual acuities in the far, intermediate and near | 1 month
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Visual acuities in the far, intermediate and near | 3 months
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Mesopic vision | 1 month
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Mesopic vision | 3 months
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Scotopic contrast sensitivity | 1 month
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.
Scotopic contrast sensitivity | 3 months
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.

SECONDARY OUTCOMES:
Spectacle independence in the far, intermediate and near | 3 months
  Spectacle independence as stated by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Bertelmann, MD, PhD, Principal Investigator — eckart.bertelmann@charite.de; Tobias Brockmann, MD, Principal Investigator — tobias.brockmann@charite.de
Locations (1):
- Charité - University Medicine Berlin, Department of Ophthalmology, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Pedrotti E, Mastropasqua R, Passilongo M, Parisi G, Marchesoni I, Marchini G. Comparison of two multifocal intraocular lens designs that differ only in near add. J Refract Surg. 2014 Nov;30(11):754-60. doi: 10.3928/1081597X-20141021-07. PMID 25375848
- [Background] Alfonso JF, Knorz M, Fernandez-Vega L, Rincon JL, Suarez E, Titke C, Kohnen T. Clinical outcomes after bilateral implantation of an apodized +3.0 D toric diffractive multifocal intraocular lens. J Cataract Refract Surg. 2014 Jan;40(1):51-9. doi: 10.1016/j.jcrs.2013.06.026. PMID 24355720
- [Background] Javitt JC, Steinert RF. Cataract extraction with multifocal intraocular lens implantation: a multinational clinical trial evaluating clinical, functional, and quality-of-life outcomes. Ophthalmology. 2000 Nov;107(11):2040-8. doi: 10.1016/s0161-6420(00)00368-7. PMID 11054329
- [Background] Vingolo EM, Grenga P, Iacobelli L, Grenga R. Visual acuity and contrast sensitivity: AcrySof ReSTOR apodized diffractive versus AcrySof SA60AT monofocal intraocular lenses. J Cataract Refract Surg. 2007 Jul;33(7):1244-7. doi: 10.1016/j.jcrs.2007.03.052. PMID 17586381
- [Background] Cillino G, Casuccio A, Pasti M, Bono V, Mencucci R, Cillino S. Working-age cataract patients: visual results, reading performance, and quality of life with three diffractive multifocal intraocular lenses. Ophthalmology. 2014 Jan;121(1):34-44. doi: 10.1016/j.ophtha.2013.06.034. Epub 2013 Aug 14. PMID 23953097
- [Background] Chiam PJ, Chan JH, Aggarwal RK, Kasaby S. ReSTOR intraocular lens implantation in cataract surgery: quality of vision. J Cataract Refract Surg. 2006 Sep;32(9):1459-63. doi: 10.1016/j.jcrs.2006.04.015. PMID 16931256